CLINICAL TRIAL: NCT04844697
Title: Exploring Resilience and Coping Strategies of Young Population in Response to Severe Acute Respiratory Syndrome Corona Virus 2 (SARS-CoV-2) Outbreak: a Longitudinal Study in a Cohort of Patients Affected by Rare Skeletal Disorders.
Brief Title: Resilience and Coping in a Rare Skeletal Disease Population to Face Coronavirus (COVID-19) Outbreak Distress: a Longitudinal Study
Acronym: RELOAD
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Luca Sangiorgi, Director of Rare Skeletal Disorders Department, Istituto Ortopedico Rizzoli
Other Study IDs: 150/2021/Oss/IOR
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Multiple Osteochondroma; Osteogenesis Imperfecta; Ollier Disease; Maffucci Syndrome
Keywords: COVID-19; Psychological Distress; e-Health; Children, Adolescents, Young Adults; Coping Strategies; Rare Diseases; Focus group
MeSH Terms: conditions — Exostoses, Multiple Hereditary; Osteogenesis Imperfecta; Enchondromatosis; COVID-19; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the COVID-19 outbreak context, people living with rare diseases have been highly troubled with anxiety, loneliness, and depression. The project evaluates resilience and coping strategies to address pandemic impact by discussion in a dedicated focus group using a web-based platform. The goal is to improve, in a sustainable manner, the coping skills and psychological well-being of children, adolescents, and young adults affected by rare skeletal diseases.

DETAILED DESCRIPTION:
March 11th, 2020, the World Health Organization (WHO) declared the SARS-CoV-2 pandemic accordingly with the spread and size of the infection.

The restrictions implemented by the governments have substantially changed people's lifestyles, facilitating the emergence of emotions such as fear, anxiety, and a sense of loneliness.

The age groups most involved by these burdens have been childhood, adolescence, and young adults. These groups have experienced dramatic changes in their daily life in order the relational, educational, and social networks. Nonetheless, these links outline the ideal environment for the development of resilience and the promotion of coping strategies to face traumatic events.

These lifestyle challenges and their consequences are even more evident in the context of the rare diseases since the outbreak containment measures have emphasized the troubles with which people affected by these conditions are daily forced to confront, in terms of access to care and treatments, resulting in increased stress and anxiety.

The current phase represents a sensitive step for the resumption of the activities in charge of the health and social service aimed at the citizens and especially to people with special needs, such as people suffering from rare diseases.

The pandemic experience has promoted new forms of meeting and contact between individuals using web-based platforms, playing a fundamental role in preserving the community and "sociality" dimensions.

In this scenario, the rare diseases could be an attractive model since the pandemic impinges over their bio-psycho-social characteristics at different levels. Resilience and coping strategies adopted by rare diseases patients could configure as an exemplum to face the psychological distress resulting from anti-pandemic measures, suggesting new approaches of taking charge by health service.

This study evaluates resilience and coping strategies to address pandemic impact by discussion in a dedicated focus group using a web-based platform. The goal is to improve, in a sustainable manner, the coping skills and psychological well-being of children, adolescents, and young adults affected by rare skeletal diseases.

ELIGIBILITY:
Inclusion Criteria:

Clinical and/or molecular diagnosis of Multiple osteochondromas; Clinical and/or molecular diagnosis of Ollier disease/Maffucci syndrome; Clinical and/or molecular diagnosis of Osteogenesis imperfecta; Consent to participate in the study

Exclusion Criteria:

Subject doesn't match the inclusion criteria

Ages: 8 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient screening and enrollment will be carried out through:
  * Rare Skeletal Disorders out-patient visit
  * Rare Skeletal Disorders in-patient visit
  * National Patients Organizations
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Resilience | Evaluation at baseline of the study
  Ego-Resiliency Scale (ER89); 14 items; 4-point Likert scale (1=does not apply at all; 2=applies slightly, if at all; 3=applies somewhat; and 4=applies very strong); Score Resiliency Trait: 47-56 Very High, 35-46 High, 23-34 Undetermined, 11-22 Low, 0-10 Very Low
Resilience | Change from baseline at 3 month
  Ego-Resiliency Scale (ER89); 14 items; 4-point Likert scale (1=does not apply at all; 2=applies slightly, if at all; 3=applies somewhat; and 4=applies very strong); Score Resiliency Trait: 47-56 Very High, 35-46 High, 23-34 Undetermined, 11-22 Low, 0-10 Very Low
Resilience | Change from baseline at 6 month
  Ego-Resiliency Scale (ER89); 14 items; 4-point Likert scale (1=does not apply at all; 2=applies slightly, if at all; 3=applies somewhat; and 4=applies very strong); Score Resiliency Trait: 47-56 Very High, 35-46 High, 23-34 Undetermined, 11-22 Low, 0-10 Very Low

SECONDARY OUTCOMES:
Anxiety | Evaluation at baseline of the study
  Hospital Anxiety and Depression Scale (HADS); 14 items: 7 items relate to anxiety and 7 relate to depression; a 4-point (0-3) Likert-scale; Cutoffs for both HADS-anxiety and HADS-depression as >= 8, and for HADS-total >= 15
Anxiety | Change from baseline at 3 month
  Hospital Anxiety and Depression Scale (HADS); 14 items: 7 items relate to anxiety and 7 relate to depression; a 4-point (0-3) Likert-scale; Cutoffs for both HADS-anxiety and HADS-depression as >= 8, and for HADS-total >= 15
Anxiety | Change from baseline at 6 month
  Hospital Anxiety and Depression Scale (HADS); 14 items: 7 items relate to anxiety and 7 relate to depression; a 4-point (0-3) Likert-scale; Cutoffs for both HADS-anxiety and HADS-depression as >= 8, and for HADS-total >= 15
Depression | Evaluation at baseline of the study
  Hospital Anxiety and Depression Scale (HADS); 14 items: 7 items relate to anxiety and 7 relate to depression; a 4-point (0-3) Likert-scale; Cutoffs for both HADS-anxiety and HADS-depression as >= 8, and for HADS-total >= 15
Depression | Change from baseline at 3 month
  Hospital Anxiety and Depression Scale (HADS); 14 items: 7 items relate to anxiety and 7 relate to depression; a 4-point (0-3) Likert-scale; Cutoffs for both HADS-anxiety and HADS-depression as >= 8, and for HADS-total >= 15
Depression | Change from baseline at 6 month
  Hospital Anxiety and Depression Scale (HADS); 14 items: 7 items relate to anxiety and 7 relate to depression; a 4-point (0-3) Likert-scale; Cutoffs for both HADS-anxiety and HADS-depression as >= 8, and for HADS-total >= 15
Loneliness | Evaluation at baseline of the study
  UCLA Loneliness Scale (Version 3); 20-item scale; 4-point rating scale (1=Never; 2=Rarely; 3=Sometimes; and 4=Often); score ranging from 20 to 80.
Loneliness | Change from baseline at 3 month
  UCLA Loneliness Scale (Version 3); UCLA Loneliness Scale (Version 3); 20-item scale; 4-point rating scale (1=Never; 2=Rarely; 3=Sometimes; and 4=Often); score ranging from 20 to 80.
Loneliness | Change from baseline at 6 month
  UCLA Loneliness Scale (Version 3); UCLA Loneliness Scale (Version 3); 20-item scale; 4-point rating scale (1=Never; 2=Rarely; 3=Sometimes; and 4=Often); score ranging from 20 to 80.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Sangiorgi, MD, Phd, Principal Investigator — IRCCS Istituto ORtopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No